CLINICAL TRIAL: NCT00610415
Title: Biopsy of Human Tumors for Cancer Stem Cell Characterization: a Feasibility Study
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: ENT0023; 98543 (Other: Stanford University Alternate IRB Approval Number); SU-12142007-934 (Other: Stanford University); NCT00610415; 10514 (Other: Stanford IRB)
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Head and Neck Cancer; Head and Neck Cancers
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples

INTERVENTIONS:
Procedure: tumor biopsy

SUMMARY:
To see if a limited sampling of tumor tissue from human subjects is a feasible way to gather adequate tissue for cancer stem cell quantification.

ELIGIBILITY:
Inclusion Criteria:1. Patients with malignant tumors seen at the Stanford University Cancer Center. Eligible patients will have a diagnosis of squamous cell carcinoma (HNSCC) and will have been seen in the Stanford Head and Neck Oncology Program. A decision to undergo surgery at Stanford will have been made, prior to recruiting patients for the study, and prior to obtaining the samples during surgery. (Histological confirmation of the diagnosis need not be made prior to obtaining consent.) 2. A definitive resection of a malignant tumor is planned. 3. Surgeon judgment that the definitive procedure will not be compromised by including

* FNA
* Core needle biopsy
* Cup forceps or punch biopsy of<4mm. 4. Informed consent documented prior to procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will have a diagnosis of squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Quantification of the cancer stem cell population by flow cytometry | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Dr. A. Dimitrios Colevas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States